CLINICAL TRIAL: NCT04609072
Title: Connect for Cancer Prevention Study: A Prospective Cohort Study Within Integrated Healthcare Systems in the US
Brief Title: Connect for Cancer Prevention Study (Connect)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000034; 000034-C
Record Dates: First submitted 2020-10-29; First posted 2020-10-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Cancer; General Research Use
Keywords: Risk Factors; medical conditions; Pathology; Blood; Urine; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Up to 200,000 men and women aged 30 to 70 years, with no personal history of cancer, and patients or members of participating integrated health care systems.

SUMMARY:
Background:

The National Cancer Institute, part of the National Institutes of Health, has partnered with nine health care systems across the U.S. to establish the Connect for Cancer Prevention Study. While researchers have made important discoveries, there is more to learn to lower the number of people affected by cancer. By taking part in Connect, participants can help researchers learn how the way we live, our genetics, and our health history may affect cancer risk.

Objective:

To study and better understand the causes of cancer and to find new ways to prevent it.

Eligibility:

The study will include 200,000 adults who get their health care from a partner health care system, are between 30 and 70 years old at enrollment, and have never had cancer. People remain eligible to join if they have or once had non-melanoma skin cancer, or a condition that may raise cancer risk (such as ductal carcinoma in situ, or DCIS).

Design:

Eligible recruits can sign up for Connect online by creating an account on MyConnect using their email address or phone number. After creating an account, they will complete the informed consent process. All information shared through MyConnect is secure to protect participant privacy. After joining the study, participants will be asked to answer online health surveys a few times a year, donate samples of blood, urine, and saliva every two to three years, and safely share access to their electronic health records with Connect. In the future, participants may donate unused samples that are collected at clinical visits, like tissue, stool, or blood, and may mail in samples collected at home. Participants may also share information from personal health trackers, like wearable devices or apps.

This information will help researchers study the health and behavior patterns that may affect cancer risk.

It takes time to understand the causes of cancer, so Connect will go on for many years. The longer people participate, the more researchers may learn. Participants can leave the study at any time.

Learn more about Connect by visiting cancer.gov/connectstudy.

DETAILED DESCRIPTION:
Study Description:

Connect is an observational cohort study that will prospectively collect exposure information and biospecimens and follow participants for cancer and other endpoints. Participants will be free of cancer at study invitation. Because most cancers develop over long periods of time and biological, behavioral and environmental factors can influence cancer development and change over time, participants will be asked to provide repeated exposure information and biological specimens. The study protocol takes advantage of developments in digital technologies as well as exposure and biomarker assessment tools to investigate suspected and emerging factors that can influence cancer development. The study data system will be built within an efficient, flexible and integrated cloud-hosted infrastructure that leverages modern interoperability standards in order to be an accessible research resource for current and future generations of scientists.

Objectives:

The primary objective is to build a state-of-the-art cohort in the US using new technologies and methods to provide a diverse and comprehensive research resource for the scientific community to study:

* cancer etiology
* precursor to tumor transformation
* cancer risk assessment
* early detection of cancer
* second cancer development and survivorship after a cancer diagnosis

The secondary objective is to establish a rich database connected to a biorepository for general research use.

Endpoints:

The primary endpoints are the continuum of cancer incidence, detection, progression, and survival. Secondary endpoints are numerous and could include methodological research, human biology, ancestry, evolution or health-related outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Due to the minimal risk nature of this protocol, all individuals interested and able to participate in Connect for Cancer Prevention, who meet the eligibility criteria at time of initial study invitation, will be able to participate. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Patients or members of participating IHCS at the time of enrollment
* Age between 30 and 70 years old at study invitation

If an individual is determined to be ineligible at the time of enrollment due to age, the individual will be allowed to re-enroll at a later time once the recruit meets the age requirement. This includes recruits that did not meet the original age requirement of 40-65 years of age but now meet the updated age range of 30-70.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria at time of initial study invitation will be excluded from participation in this study:

* Individuals with a confirmed history of invasive cancer (other than non-melanoma skin cancer)
* Individuals with known cognitive impairment documented in their medical record

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients or members of participating health care organizations around the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2070-12-31 (Estimated); Study Completion 2070-12-31 (Estimated)

PRIMARY OUTCOMES:
cancer incidence, progression, and mortality | year one and onward
  cancer incidence, progression, and mortality outcomes could include, but are not limited to:early biological effects (e.g., inflammation or metabolomic markers) related to cancer, intermediate biomarkers, cancer precursors, cancer risk factors, cancer incidence, cause of death, cancer survival, risk of second cancers and survivorship

SECONDARY OUTCOMES:
general research use | year zero and onward
  The endpoints are limitless and could include methodological research, human biology, ancestry, evolution or health-related outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas A Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (10):
- United States (10):
  - Kaiser Permanente Colorado, Denver, Colorado
  - Kaiser Permanente Georgia, Atlanta, Georgia
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - Henry Ford Health Systems, Detroit, Michigan
  - HealthPartners, Minneapolis, Minnesota
  - Kaiser Permanente Northwest, Portland, Oregon
  - Sanford Health, Sioux Falls, South Dakota
  - Baylor Scott and White Health, Dallas, Texas
  - Marshfield Clinic Health System, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All collected Connect IPD will be provided to the scientific community following the governance principles outlined in the protocol.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting in 2023
Access Criteria: Please see Sections 8 and 9.11 of the protocol that address data sharing.

REFERENCES:
- [Background] Rebbeck TR, Burns-White K, Chan AT, Emmons K, Freedman M, Hunter DJ, Kraft P, Laden F, Mucci L, Parmigiani G, Schrag D, Syngal S, Tamimi RM, Viswanath K, Yurgelun MB, Garber JE. Precision Prevention and Early Detection of Cancer: Fundamental Principles. Cancer Discov. 2018 Jul;8(7):803-811. doi: 10.1158/2159-8290.CD-17-1415. Epub 2018 Jun 15. PMID 29907587
- See also: https://www.cancer.gov/connect-prevention-study/ — https://www.cancer.gov/connect-prevention-study/